CLINICAL TRIAL: NCT02469597
Title: Single Dose of Furosemide to Improve Respiratory Distress in Moderate to Severe Bronchiolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Sandeep Gangadharan, Principal Investigator, MD, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-260B
Record Dates: First submitted 2015-05-24; First posted 2015-06-11 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-06

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Dose of Furosemide (Experimental): Furosemide 1 dose
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): Normal saline 1 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Furosemide — 1 mg/kg intravenous or oral (will give oral unless patient has peripheral IV access in place), maximum dose 10mg (1ml), x 1 dose
  Other Names: Lasix
  Arms: Single Dose of Furosemide
Drug: Placebo — 0.1ml/kg intravenous or oral (Normal Saline) (will give oral unless patient has peripheral IV access in place), maximum dose 1ml, x 1 dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if administration of an early single dose of a diuretic (furosemide) to children with moderate to severe bronchiolitis can reduce extravascular lung water in an effort to reduce respiratory rate, retractions, intubations, and length of stay.

DETAILED DESCRIPTION:
Randomization and Blinding:

Subjects will be randomly assigned by a 1:1 ratio to either furosemide or placebo. The Biostatistics Unit will develop a randomization procedure using a permuted block design. The randomization will be stratified by mode of delivery of furosemide: IV or PO. Blinding will be maintained at all times throughout the study. The only unblinded study personnel will be the pharmacy department who will dispense either of placebo or furosemide to each patient. Blinding will be broken only in the case of allergic reaction in which case a pediatric attending physician, not involved with the study (designated prior to study initiation) will be notified to access the intervention of that patient. If such an event should occur, the primary investigator and IRB will be notified by e-mail/phone, and an adverse event will be documented.

Materials / Methods:

All patients aged 0-4 years old with primary diagnosis of bronchiolitis on assessment by the Emergency Department will be evaluated for inclusion to study. The goal patient enrollment is 100 patients, which is required to achieve statistical significance (see below). As this study focuses on moderate (admitted) to severe (requiring mechanical ventilation) patients with bronchiolitis, further documentation would be completed on a data collection sheet. Randomization will occur upon consent to study. In collaboration with the Biostatistics Unit, patients will be randomly assigned by a 1:1 ratio to either furosemide or placebo. There will be a randomization procedure using a permuted block design. The randomization will be stratified by mode of delivery of intervention: IV or PO. The corresponding intervention (placebo or furosemide) will then be dispensed by pharmacy for administration in a blinded manner by the patient's nurse and/or physician. Either a single dose furosemide (1mg/kg or 10mg - whichever is less) will be administered orally PO (or intravenously [IV] if IV is present), or a placebo of equal volume. Ideally, the intervention dose will be administered as early as possible (immediately after decision to admit was made and consent obtained). Subsequent retrieval of that data will be done by study personnel. Data recorded on the data collection sheet can include: O2 Saturation/Weight (pre-intervention and, 2 and 4 hours post-furosemide/control), Age, Gender, Prematurity (<32 weeks gestation), history of mechanical ventilation, history of wheeze / asthma, history of furosemide use, interventions prior to furosemide (racemic epinephrine, albuterol, or non-invasive ventilation), RSV / Influenza status, degree of dehydration (mild / moderate / severe), onset of symptoms prior to triage, +/- apnea, timing from initiation of visit until furosemide administration and/or non-invasive/invasive ventilator support, and reason for admission to ICU if necessary.

Considerations for all analyses:

All analyses will be carried out under the intention to treat principle; patients will be analyzed according to the groups to which they were randomized. (However, it is likely that the intention to treat population will be the same as the per protocol population.)

The primary analyses will be carried out for all patients. Mode of delivery of furosemide (IV vs. PO) will not be included in the analysis, as the aim of the study is to examine the effects of furosemide, regardless of mode of delivery. Randomization will be stratified by mode of delivery, so that the distribution of mode of delivery will be the same for the two treatment groups. Secondary subgroup analyses will be performed analyzing each mode of delivery (IV, PO), separately. These secondary subgroup analyses will be the same as the primary analyses.

Analyses for Specific Aims:

1. The association between treatment (furosemide) and control (placebo) groups will be compared using the chi-square test for the categorical outcomes (25% decrease in respiratory rate, intubation, etc).

Percent change in respiratory rate will be compared using the two sample t-test. If the usual assumptions required for the t-test are not met, then either a suitable transformation, or an appropriate non-parametric test (the Mann-Whitney test), will be used.

Length of stay (LOS) will be compared using the Mann-Whitney test. In the event that not all participants are followed until discharge from the hospital (in-hospital mortality, not discharged by end of study period), survival methods will be used (LOS will be estimated using the product-limit method, and the treatment groups will be compared using the log-rank test).

Sample Size Justification:

Based on clinical experience, we believe that very few patients who are admitted with bronchiolitis will have a response (as described in the primary outcome: a decrease in respiratory rate of 25% or more, or a return to their age appropriate respiration rate), at 2 hours post administration of placebo. To be conservative, it is assumed that the response to placebo will be no higher than 5%. It is believed that a clinically meaningful response rate would be 25% of patients at 2 hours after administration of furosemide. The proposed sample size of 49 subjects per group will yield 80% power to detect such a difference using a chi-square test with a 0.05 significance level.

Clinical Outcomes Justification:

Given the transient nature of bronchiolitis, as symptoms typically peak treatment is sought. Along with furosemide's half life of approximately 6hrs, there could be a correlation drawn between those children intubated (respiratory failure) or not, as it relates to when furosemide was given. Twenty-four hours is a reasonable observation period to correlate to the intervention. Intubation beyond that time point may infer that similar treatments of furosemide were warranted given the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Bronchiolitis
* Admission required per Emergency Department Physician

Exclusion Criteria:

* No legal guardian present
* Sulfa allergy
* Patient currently on existing diuretic therapy
* Tracheostomy
* Mild respiratory distress (not requiring admission)
* Hypotension / Hemodynamic Instability (defined by age specific criteria at time of intervention)
* Supplemental Oxygen at home
* History of Dialysis / Renal Disease
* Those enrolled in another drug interventional study

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Gangadharan, MD, Principal Investigator — Northwell Health
Locations (1):
- Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

REFERENCES:
- [Background] Pelletier AJ, Mansbach JM, Camargo CA Jr. Direct medical costs of bronchiolitis hospitalizations in the United States. Pediatrics. 2006 Dec;118(6):2418-23. doi: 10.1542/peds.2006-1193. PMID 17142527
- [Background] Baker MD. Pitfalls in the use of clinical asthma scoring. Am J Dis Child. 1988 Feb;142(2):183-5. doi: 10.1001/archpedi.1988.02150020085035. PMID 3341321
- [Background] Farias JA, Fernandez A, Monteverde E, Flores JC, Baltodano A, Menchaca A, Poterala R, Panico F, Johnson M, von Dessauer B, Donoso A, Zavala I, Zavala C, Troster E, Pena Y, Flamenco C, Almeida H, Nilda V, Esteban A; Latin-American Group for Mechanical Ventilation in Children. Mechanical ventilation in pediatric intensive care units during the season for acute lower respiratory infection: a multicenter study. Pediatr Crit Care Med. 2012 Mar;13(2):158-64. doi: 10.1097/PCC.0b013e3182257b82. PMID 21725275
- [Background] Hernando Puente M, Lopez-Herce Cid J, Bellon Cano JM, Villaescusa JU, Santiago Lozano MJ, Sanchez Galindo A. [Prognostic factors for bronchiolitis complications in a pediatric intensive care unit]. An Pediatr (Barc). 2009 Jan;70(1):27-33. doi: 10.1016/j.anpedi.2008.08.004. Epub 2008 Nov 25. Spanish. PMID 19174116
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Rush MG, Engelhardt B, Parker RA, Hazinski TA. Double-blind, placebo-controlled trial of alternate-day furosemide therapy in infants with chronic bronchopulmonary dysplasia. J Pediatr. 1990 Jul;117(1 Pt 1):112-8. doi: 10.1016/s0022-3476(05)82458-8. PMID 2196353
- [Background] Stewart A, Brion LP. Intravenous or enteral loop diuretics for preterm infants with (or developing) chronic lung disease. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD001453. doi: 10.1002/14651858.CD001453.pub2. PMID 21901676
- [Background] Hagadorn JI, Sanders MR, Staves C, Herson VC, Daigle K. Diuretics for very low birth weight infants in the first 28 days: a survey of the U.S. neonatologists. J Perinatol. 2011 Oct;31(10):677-81. doi: 10.1038/jp.2011.11. Epub 2011 Mar 10. PMID 21394079
- [Background] Green TP. The pharmacologic basis of diuretic therapy in the newborn. Clin Perinatol. 1987 Dec;14(4):951-64. PMID 3322632
- [Background] Hufnagle KG, Khan SN, Penn D, Cacciarelli A, Williams P. Renal calcifications: a complication of long-term furosemide therapy in preterm infants. Pediatrics. 1982 Sep;70(3):360-3. PMID 7110808
- [Background] Ross BS, Pollak A, Oh W. The pharmacologic effects of furosemide therapy in the low-birth-weight infant. J Pediatr. 1978 Jan;92(1):149-52. doi: 10.1016/s0022-3476(78)80098-5. PMID 22591
- [Background] Ghanekar AG, Das Gupta V, Gibbs CW Jr. Stability of furosemide in aqueous systems. J Pharm Sci. 1978 Jun;67(6):808-11. doi: 10.1002/jps.2600670621. PMID 660463
- [Derived] Williamson K, Bredin G, Avarello J, Gangadharan S. A Randomized Controlled Trial of a Single Dose Furosemide to Improve Respiratory Distress in Moderate to Severe Bronchiolitis. J Emerg Med. 2018 Jan;54(1):40-46. doi: 10.1016/j.jemermed.2017.08.099. Epub 2017 Nov 23. PMID 29174754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at a tertiary care, academic children's hospital in the Pediatric Emergency Department from February 2013 to March 2016.
Period: Overall Study
Arm/Group | Single Dose of Furosemide | Placebo
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose of Furosemide | Placebo | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 24 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.7 (5.5) | 8.1 (6.8) | 7.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Rate
Time Frame: 2 hours after medication adminstration
Measure: Least Squares Mean (Standard Error); unit: Percentage change in respiratory rate
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
Percentage change in respiratory rate | -3.7 (5.5) | -1.7 (5.3)

2. Primary Outcome: Respiratory Rate
Time Frame: 4 hours after medication adminstration
Measure: Least Squares Mean (Standard Error); unit: Percentage change in respiratory rate
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
Percentage change in respiratory rate | -2.8 (6.5) | -5.4 (6.3)

3. Primary Outcome: Oxygen Saturation
Time Frame: 2 hours after medication adminstration
Measure: Least Squares Mean (Standard Error); unit: Percentage change in oxygen saturation
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
Percentage change in oxygen saturation | -0.14 (0.67) | 0.2 (0.6)

4. Primary Outcome: Oxygen Saturation
Time Frame: 4 hours after medication adminstration
Measure: Least Squares Mean (Standard Error); unit: Percentage change in oxygen saturation
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
Percentage change in oxygen saturation | -0.19 (0.58) | 0.29 (0.84)

5. Secondary Outcome: Patient Needing Endotracheal Intubation
Time Frame: Within 72 hours of medication administration
Measure: Number; unit: participants
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
participants | 0 | 0

6. Secondary Outcome: Length of Hospital Stay
Time Frame: Participants will be followed for the duration of hospital stay up to 1 week
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Single Dose of Furosemide | Placebo
Number analyzed (Participants) | 22 | 24
Days | 3.1 (0.5) | 3.0 (0.5)

ADVERSE EVENTS:
Arm/Group | Single Dose of Furosemide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

LIMITATIONS AND CAVEATS:
The trial was ended early due to recruitment difficulties.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes